CLINICAL TRIAL: NCT04280718
Title: Open-label Extension of the ARGX-113-1802 Trial to Investigate the Long-term Safety, Tolerability, and Efficacy of Efgartigimod PH20 SC in Patients With Chronic Inflammatory Demyelinating Polyneuropathy (CIDP)
Brief Title: A Study to Assess the Long-term Safety and Efficacy of a Subcutaneous Formulation of Efgartigimod in Adults With Chronic Inflammatory Demyelinating Polyneuropathy (CIDP, an Autoimmune Disorder That Affects the Peripheral Nerves)
Acronym: ADHERE+
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: argenx (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ARGX-113-1902; 2019-003107-35 (EudraCT Number)
Record Dates: First submitted 2020-02-20; First posted 2020-02-21 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Chronic Inflammatory Demyelinating Polyneuropathy (CIDP)
MeSH Terms: conditions — Polyradiculoneuropathy, Chronic Inflammatory Demyelinating | interventions — efgartigimod alfa

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- efgartigimod PH20 SC (Experimental): Patients treated with efgartigimod PH20 SC
  Interventions: Biological: Efgartigimod PH20 SC

INTERVENTIONS:
Biological: Efgartigimod PH20 SC — Subcutaneous administration of efgartigimod
  Other Names: ARGX-113

SUMMARY:
This is the open-label extension study of phase II ARGX-113-1802 to evaluate the long-term safety and efficacy of the subcutaneous formulation of efgartigimod in adults with CIDP.

Patients already stabilized on efgartigimod PH20 SC will also have the opportunity to participate in a sub study to explore less frequent dosing of efgartigimod PH20 SC.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to understand the requirements of the trial, provide written informed consent (including consent for the use and disclosure of research-related health information), willingness and ability to comply with the trial protocol procedures (including required trial visits) of this trial.
2. Male or female patient with one of the following options:

   * Have completed the Week-48 visit of Stage B of the ARGX-113-1802 trial and are considered to be eligible for treatment with efgartigimod PH20 SC; or
   * Have deteriorated during Stage B of the ARGX-113-1802 trial and are considered to be eligible for treatment with efgartigimod PH20 SC, or
   * Have been offered the participation in the OLE trial due to early termination of the ARGX-113-1802 trial (because sufficient events for the primary endpoint analysis of the that trial have been reached and it is stopped) and are considered to be eligible for treatment with efgartigimod PH20 SC treatment; or
   * Have completed the Week-48 visit of the previous cycle of the OLE trial and are considered to be eligible to continue with efgartigimod PH20 SC treatment.
3. Women of childbearing potential who have a negative urine pregnancy test at baseline before IMP administration.
4. Women of childbearing potential must use an acceptable method of contraception from signing the ICF until the date of the last administration of IMP.

Exclusion Criteria:

1. Week-48/ED visit in the ARGX-113-1802 trial or the Week-48 visit of the previous OLE participation occurred more than 14 days prior to SD1 of the OLE trial or the start of a new treatment cycle in the OLE trial and more than 21 days since the last dose of IMP.
2. Pregnant and lactating women and those intending to become pregnant during the trial.
3. Patients with clinical evidence of other significant serious disease or patients who underwent a recent or have a planned major surgery, or patients who (intend to) use prohibited medications (see protocol) and therapies during the trial, or any other reason which could confound the results of the trial or put the patient at undue risk.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 229 (Actual)
Dates: Start 2020-09-18 (Actual); Primary Completion 2027-04-30 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events and serious adverse events | Up to 48 weeks per cycle (each cycle is 48 weeks) until the end of the study

SECONDARY OUTCOMES:
Change from baseline over time of the adjusted INCAT score | Up to 48 weeks per cycle (each cycle is 48 weeks) until the end of the study
  The Adjusted Inflammatory Neuropathy Cause and Treatment Disability Score (aINCAT) score is a 10-point scale that covers the functionality of legs and arms. The score varies between 0 and 10 (higher score, worse outcome).
Change from baseline over time of the MRC Sum score | Up to 48 weeks per cycle (each cycle is 48 weeks) until the end of the study
  The Medical Research Council Sum Score evaluates motor strength. Evaluated on 6 muscle groups on each side, the score varies from 0 to 60 (lower score, worse outcome).
Change from baseline over time of I-RODS disability scores | Up to 48 weeks per cycle (each cycle is 48 weeks) until the end of the study
  Inflammatory Rasch-built Overall Disability Scale (I-RODS) assesses the limitations of activities and social participation in patients with inflammatory neuropathies like CIDP. The score ranges from 0 to 100 (higher score, worse outcome).
Change from baseline over time of mean grip strength | Up to 48 weeks per cycle (each cycle is 48 weeks) until the end of the study
Change from baseline over time of TUG score | Up to 48 weeks per cycle (each cycle is 48 weeks) until the end of the study
  The Timed Up and Go Test (TUG) is a simple test to assess a person's mobility in which the time expended to rise from a chair, walk 3 meters, turn around, walk back to the chair, and sit down is measured.
Percentage of patients without clinical deterioration over time, defined by adjusted INCAT deterioration ≥1 point compared to baseline. | Up to 48 weeks per cycle (each cycle is 48 weeks) until the end of the study
  The Adjusted Inflammatory Neuropathy Cause and Treatment Disability Score (aINCAT) score is a 10-point scale that covers the functionality of legs and arms. The score varies between 0 and 10 (higher score, worse outcome).
Percentage of patients with titers of binding antibodies towards efgartigimod and the presence of neutralizing antibodies against efgartigimod. | Up to 51 weeks
Efgartigimod serum concentrations | Up to 51 weeks
Changes from baseline over time of serum IgG levels (total) | Up to 48 weeks per cycle (each cycle is 48 weeks) until the end of the study
Change from baseline over time in EQ-5D-5L | Up to 48 weeks per cycle (each cycle is 48 weeks) until the end of the study
  EQ-5D-5L questionnaire is a patient-reported outcome measure, ranging 0 to 100 (lower score, worse outcome).
Change from baseline over time in BPI SF | Up to 48 weeks per cycle (each cycle is 48 weeks) until the end of the study
  The Brief Pain Inventory-Short Form (BPI-SF) is a patient-reported outcome measure to assess pain severity and pain interference
Change from baseline over time in TSQM-9 | Up to 48 weeks per cycle (each cycle is 48 weeks) until the end of the study
  The Treatment Satisfaction Questionnaire for Medication (TSQM) is a 9-item questionnaire to assess treatment satisfaction in naturalistic study designs, in which there is potential that the administration of the side effects domain of the TSQM would interfere with routine clinical care
Change from baseline over time in RT-FSS | Up to 48 weeks per cycle (each cycle is 48 weeks) until the end of the study
  The Rasch-Transformed Fatigue Severity Scale (RT-FSS) is a 7-item self-reported questionnaire designed to differentiate fatigue from clinical depression. The participant has to rate from 0 to 3 their level of fatigue on 7 items (low score indicates that the statement is not very appropriate, and high score indicates agreement).
Change from baseline over time in HADS | Up to 48 weeks per cycle (each cycle is 48 weeks) until the end of the study
  The Hospital Anxiety and Depression Scale (HADS) aims to measure symptoms of anxiety and depression in people with physical health problems. HADS is a 14-item scale with 7 items related to anxiety and 7 to depression
Percentage of patients performing self-administration over time | Up to 48 weeks per cycle (each cycle is 48 weeks) until the end of the study
Percentage of patients with treatment administered by caregiver over time. | Up to 48 weeks per cycle (each cycle is 48 weeks) until the end of the study

CONTACTS AND LOCATIONS:
Locations (147):
- United States (25):
  - Investigator site 0010065, Birmingham, Alabama
  - Investigator site 0010013, Phoenix, Arizona
  - Investigator site 0010055, Scottsdale, Arizona
  - Investigator site 0010032, Carlsbad, California
  - Investigator site 10190, Pomona, California
  - Investigator site 0010160, Rancho Mirage, California
  - Investigator site 0010071, San Francisco, California
  - Investigator site 0010057, Centennial, Colorado
  - Investigator site 0010072, Boca Raton, Florida
  - Investigator site 0010144, Coral Springs, Florida
  - Investigator site 0010023, Jacksonville, Florida
  - Investigator site 0010068, Maitland, Florida
  - Investigator site 0010059, Miami, Florida
  - Investigator site 0010006, Tampa, Florida
  - Investigator site 0010011, Iowa City, Iowa
  - Investigator site 0010015, Fairway, Kansas
  - Investigator site 10147, Lexington, Kentucky
  - Investigator site 10168, New York, New York
  - Investigator site 0010003, Chapel Hill, North Carolina
  - Investigator site 0010064, Columbus, Ohio
  - Investigator site 0010007, Philadelphia, Pennsylvania
  - Investigator site 0010047, Philadelphia, Pennsylvania
  - Investigator Site 0010066, Austin, Texas
  - Investigator site 0010009, San Antonio, Texas
  - Investigator site 0010061, Richmond, Virginia
- Austria (3):
  - Investigator site 0430007, Innsbruck
  - Investigator site 0430008, Linz
  - Investigator site 0430005, Vienna
- Belgium (4):
  - Investigator site 0320016, Edegem
  - Investigator site 0320009, Leuven
  - Investigator site 320024, Liège
  - Investigator site 320022, Woluwe-Saint-Lambert
- Bulgaria (4):
  - Investigator site 3590007, Pleven
  - Investigator site 3590005, Sofia
  - Investigator site 3590008, Sofia
  - Investigator site 3590006, Sofia
- China (19):
  - Investigator site 0860033, Beijing
  - Investigator site 860041, Changsha
  - Investigator site 0860036, Chengdu
  - Investigator site 860049, Chifeng
  - Investigator site 0860038, Fuzhou
  - Investigator site 0860050, Guangzhou
  - Investigator site 0860032, Guanzhou
  - Investigator site 0860045, Guiyang
  - Investigator site 0860035, Hangzhou
  - Investigator site 0860031, Jinan
  - Investigator site 0860040, Nanchang
  - Investigator site 0860043, Nanjing
  - Investigator site 0860028, Shanghai
  - Investigator site 860047, Shanghai
  - Investigator site 0860042, Tianjin
  - Investigator site 0860034, Wuhan
  - Investigator site 0860029, Wuhan
  - Investigator site 0860048, Xi'an
  - Investigator site 0860054, Xianyang
- Investigator site 4200010, Hradec Králové, Czechia
- Denmark (3):
  - Investigator site 0450002, Aarhus
  - Investigator site 0450001, Copenhagen
  - Investigator site 0450003, Odense
- France (9):
  - Investigator site 00330034, Angers
  - Investigator site 0330013, Bordeaux
  - Investigator site 330033, Clermont-Ferrand
  - Investigator site 0330023, Le Kremlin-Bicêtre
  - Investigator site 0330024, Limoges
  - Investigator site 330022, Nantes
  - Investigator site 0330021, Nice
  - Investigator site 0330035, Paris
  - Investigator site 0330020, Strasbourg
- Georgia (5):
  - Investigator site 9950020, Kutaisi
  - Investigator site 9950004, Tbilisi
  - Investigator site 9950005, Tbilisi
  - Investigator site 9950002, Tbilisi
  - Investigator Site 9950003, Tbilisi
- Germany (6):
  - Investigator site 490044, Bochum
  - Investigator site 0490013, Cologne
  - Investigator site 490045, Essen
  - Investigator site 490021, Göttingen
  - Investigator site 0490016, Kiel
  - Investigator site 0490019, Potsdam
- Investigator site 9720004, Tel Aviv, Israel
- Italy (9):
  - Investigator site 0390022, Brescia
  - Investigator site 390029, Florence
  - Investigator site 0390024, Genova
  - Investigator site 390027, Messina
  - Investigator site 0390003, Milan
  - Investigator site 0390026, Milan
  - Investigator site 0390023, Pisa
  - Investigator site 0390008, Roma
  - Investigator site 0390042, Torino
- Japan (18):
  - Investigator site 0810035, Bunkyō City
  - Investigator site 0810002, Chiba
  - Investigator site 0810030, Fuchū
  - Investigator site 0810031, Fukuoka
  - Investigator site 0810065, Ginowan
  - Investigator site 0810066, Hakodate
  - Investigator site 0810058, Hiroshima
  - Investigator site 0810029, Kawagoe
  - Investigator site 0810026, Kodaira
  - Investigator site 810061, Kyoto
  - Investigator site 0810027, Mibu
  - Investigator site 0810032, Nagoya
  - Investigator site 0810003, Osaka
  - Investigator site 0810007, Osaka
  - Investigator site 0810063, Suita
  - Investigator site 0810036, tabashi City
  - Investigator site 0810064, Tokushima
  - Investigator site 0810060, Yokohama
- Investigator site 31, Riga, Latvia
- Netherlands (2):
  - Investigator site 0310010, Amsterdam
  - Investigator site 0310011, Rotterdam
- Poland (5):
  - Investigator site 0480024, Krakow
  - Investigator site 0480018, Krakow
  - Investigator site 0480020, Lodz
  - Investigator Site 0480017, Lublin
  - Investigator site 0480022, Warsaw
- Romania (4):
  - Investigator site 040002, Brasov
  - Investigator site 040001, Bucharest
  - Investigator site 040004, Constanța
  - Investigator site 040003, Timișoara
- Russia (7):
  - Investigator site 070017, Kazan'
  - Investigator site 0070023, Kazan'
  - Investigator site 0070020, Moscow
  - Investigator site 70021, Moscow
  - Investigator site 0070019, Rostov-on-Don
  - Investigator site 0070014, Saint Petersburg
  - Investigator site 0070021, Saransk
- Serbia (3):
  - Investigator site 3810001, Belgrade
  - Investigator site 3810003, Belgrade
  - Investigator site 3810004, Kragujevac
- Spain (3):
  - Investigator site 0340021, Badalona
  - Investigator site 0340038, Barcelona
  - Investigator site 0340018, Madrid
- Taiwan (4):
  - Investigator site 8860013, Tainan
  - Investigator site 8860012, Taipei
  - Investigator site 8860016, Taipei
  - Investigator site 8860017, Taoyuan District
- Turkey (Türkiye) (3):
  - Investigator site 900025, Bursa
  - Investigator site 900021, Izmir
  - Investigator site 900022, Samsun
- Ukraine (5):
  - Investigator Site 3800012, Dnipro
  - Investigator Site 3800010, Ivano-Frankivsk
  - Investigator site 3100013, Kyiv
  - Investigator site 3800008, Lutsk
  - Investigator site 3800011, Zaporizhzhya
- United Kingdom (3):
  - Investigator site 440026, London
  - Investigator site 0440016, Oxford
  - Investigator site 0440018, Sheffield

IPD SHARING:
Plan to Share IPD: Undecided